CLINICAL TRIAL: NCT03408600
Title: Physiologic Indicators for Prognosis in Abdominal Sepsis (PIPAS) Study
Brief Title: Physiologic Indicators for Prognosis in Abdominal Sepsis Study
Acronym: PIPAS
Status: Completed | Type: Observational
Sponsor: World Society of Emergency Surgery (Other)
Responsible Party: Principal Investigator, Massimo Sartelli, Director, World Society of Emergency Surgery
Other Study IDs: WSES/4
Record Dates: First submitted 2018-01-05; First posted 2018-01-24 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-01

CONDITIONS: Acute Peritonitis; Abdominal Sepsis
Keywords: Abdominal sepsis; Secondary peritonitis; Complicated intra-abdominal infections
MeSH Terms: conditions — Intraabdominal Infections; Peritonitis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Management — To evaluate vital signs in a global cohort of patients with acute peritonitis, determining which parameters are statistically significant to predict in-hospital mortality and ICU admission.

SUMMARY:
Early detection and timely therapeutic intervention can improve the prognosis of patients with sepsis. However, early diagnosis of sepsis can be difficult; because determining which patients presenting with signs of infection during an initial evaluation, do currently have, or will later develop a more serious illness is not easy.

Physiological deterioration often precedes clinical deterioration as patients develop critical illness. In this study, the investigators aim to evaluate vital signs in a global cohort of patients with acute secondary peritonitis, determining which parameters are statistically significant to predict in-hospital mortality and ICU admission.

DETAILED DESCRIPTION:
The study will be a worldwide multicenter observational study. The study will include patients admitted in the surgical department with acute peritonitis during a four-month study period (February 1, 2018 - May 31, 2018).

The study will not attempt to change or modify the clinical practice of the participating physicians: neither informed consent or formal approval by local Ethics Committee will be required because of the purely observational nature of the study.

The study will be monitored by the principal investigator, which will investigate and verify missing or unclear data submitted to a central database.

The study protocol has been approved by the board of the WSES and the study will be conducted under its supervision. The board of the WSES grants the proper ethical conduct of the study.

The data collection will be anonymous, as well as the name of the patients or hospital will be not collected in the website. Every hospital will continue following their ethical standards and local rules. The list of the submitted cases will not be recognized by investigators and linked to the submitting hospital. Individual researchers will take personal responsibility of data collection of this study.

In each center, the coordinator will collect and fill the data in an online case report system. These data included the following:

* Patient and disease characteristics
* Diagnostic profiles
* Treatment profiles
* Post-operative course

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of acute (secondary) localized or diffuse peritonitis.

Exclusion Criteria:

- Clinical diagnosis of acute pancreatitis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to surgical departments with acute secondary peritonitis
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Respiratory rate predicting mortality in patients with acute secondary peritonitis at admission | 24 weeks
  Respiratory rate (breaths/min);
Blood oxygen saturation level predicting mortality in patients with acute secondary peritonitis at admission | 24 weeks
  Blood oxygen saturation level (SpO2) (%) in air
Core temperature predicting mortality in patients with acute secondary peritonitis at admission | 24 weeks
  Core temperature (°C);
Systolic blood pressure predicting mortality in patients with acute secondary peritonitis at admission | 24 weeks
  Systolic blood pressure (mmHg);
Hearth rate predicting mortality in patients with acute secondary peritonitis at admission | 24 weeks
  Hearth rate (bpm);
Responsiveness predicting mortality in patients with acute secondary peritonitis at admission | 24 weeks
  Alert/verbal/painful/unresponsive (AVPU) responsiveness scale;

CONTACTS AND LOCATIONS:
Locations (1):
- WSES, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes